CLINICAL TRIAL: NCT00906737
Title: Targeted Lower Extremity Joint Training Effects on MS Gait Abnormalities
Brief Title: Effects of Targeted Lower Extremity Joint Training on Multiple Sclerosis (MS) Gait Abnormalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Jennifer Fawcett, Research Manager, Mount Sinai Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AL0002
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Gait; foot-drop; Ankle-Bot; Physical Therapy; Gait Abnormalities
MeSH Terms: conditions — Multiple Sclerosis; Peroneal Neuropathies; Mobility Limitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ankle-Bot Training (Experimental): Subjects in this group receive focused ankle training using the ankle-bot device.
  Interventions: Device: Ankle-bot
- Conventional Therapy (Active Comparator): Subjects in this group will receive conventional focused ankle physical therapy.
  Interventions: Other: Conventional focused ankle therapy
- Control (No Intervention): Subjects in this group will not receive treatment; they will continue their usual care.

INTERVENTIONS:
Device: Ankle-bot — The Ankle-bot is a piece of robotic therapy equipment for the ankle. In this study, it will be used to guide and assist the subject into ankle flexion, extension, inversion and eversion.
  Arms: Ankle-Bot Training
Other: Conventional focused ankle therapy — Conventional focused ankle therapy will be performed by a physical therapist.
  Arms: Conventional Therapy

SUMMARY:
This study is being done to test the possible benefits of task-specific focused ankle training using the Ankle-Bot on subjects with Multiple Sclerosis who have "foot-drop." The study also compares the effectiveness of task-specific focused ankle training using the Ankle-Bot with conventional focused ankle therapy in improving the gait of subjects with MS.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of MS
* EDSS level between 3.5 - 6.0
* Unilateral foot-drop
* Able to ambulate 25 ft. with no more than a unilateral assistive device

Exclusion Criteria:

* Lower extremity injuries that limit range of motion or function
* Unable to demonstrate an understanding of the process of the study and/or fully understand instructions in order to safely participate in the study and use study equipment
* Unable to fit safely and properly into the Ankle-Bot device

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Gait Parameters | Baseline, throughout study enrollment, and at 1 month and 3 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Albert Lo, M.D., Ph. D., Principal Investigator — Mandell Center for Multiple Sclerosis at Mount Sinai Rehabilitation Hospital
Locations (1):
- Mandell Center for Multiple Sclerosis at Mount Sinai Rehabilitation Hospital, Hartford, Connecticut, United States

REFERENCES:
- See also: Mandell Center for Multiple Sclerosis home page — http://www.saintfrancisdoctors.com/ms/